CLINICAL TRIAL: NCT06461273
Title: Food is Medicine vs Lifestyle Medicine: A Community Based Pragmatic Randomized Control Trial for Patients With Cardiovascular Kidney Metabolic (CKM) Syndrome
Brief Title: Food is Medicine vs Lifestyle Medicine For Cardiovascular Kidney Metabolic (CKM) Syndrome
Acronym: FiLMED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Ethos Farm to Health (Unknown)
Responsible Party: Principal Investigator, Andrew D. Lynch, PT, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2024000459
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus; Metabolic Syndrome; Obesity; Hypertension,Essential; Hyperlipidemias; Cardiovascular Diseases; Kidney Disease, Chronic
Keywords: Lifestyle Medicine; Food Is Medicine; Metabolic Syndrome; Lifestyle Related Diseases; Cardiovascular diseases; Type 2 Diabetes; Cardiovascular Kidney Metabolic Syndrome; Dietary Modification; Exercise; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome; Obesity; Essential Hypertension; Hyperlipidemias; Cardiovascular Diseases; Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle Medicine (Experimental): 20 Patients will participate in a lifestyle medicine program that includes activities and lessons in urban agriculture, nutrition education, culinary education, and exercise with a team that includes a chef, physician, farmer, and physical therapist.
  This group will meet one day per week for a 3-hour period for a total of 12-weeks.
  Interventions: Behavioral: Lifestyle Medicine Program
- Food is Medicine (Active Comparator): As a comparison group, 20 patients will be randomized to participate in a 12-week medically tailored grocery program.
  Interventions: Behavioral: Medically Tailored Groceries
- Usual Care (No Intervention): The usual care arm will serve as the control group with a total of 20 patients. The control arm will undergo the standard of care and continue their current treatment plan as coordinated with their primary care physician throughout the course of the study.

INTERVENTIONS:
Behavioral: Lifestyle Medicine Program — Participants will engage in culinary and nutrition education for 6 weeks curated by a professional chef working in conjunction with the project team from community partner Ethos Farm to Health. Lessons will be adapted from the American College of Lifestyle Medicine (ACLM) Culinary Medicine Curriculum
  Participants will engage in exercise sessions on weeks without culinary and nutrition instruction for a total of 6 weeks. Exercise sessions will include a variety of activities to include calisthenics, weight training, walking, running, dance, and games delivered by the Rutgers physical therapy team.
  Urban Agriculture lessons will occur longitudinally throughout the 12-week course. Participants will learn to cultivate a variety of crops in limited spaces, emphasizing sustainable practices and the importance of local food systems in urban communities.
  Additionally, this arm will receive a supplemental food box weekly consistent with the dietary pattern set forth by ACLM.
  Arms: Lifestyle Medicine
Behavioral: Medically Tailored Groceries — Participants in the "Food is Medicine" arm will receive a supplemental food box weekly curated by a registered dietician and dietetics students. Each food box will contain seasonally available fruit and vegetables and other items including protein, dairy/cheese, and legumes that may be available at the time of the food box delivery. Each box will contain approximately 8 pounds of food and all participants in this group will receive the same food items. Classes and educational materials provided will be tailored to the specific foods contained in the weekly food box and will include simple preparation methods, recipes, nutrition information and grocery shopping tips.
  Arms: Food is Medicine

SUMMARY:
The investigators are piloting a 3 month community-based lifestyle medicine program that incorporates experiences and education in urban agriculture, nutrition, culinary arts, and physical fitness to test the hypothesis whether this improves clinical and socio-behavioral outcomes of participants with Cardiovascular Kidney Metabolic (CKM) syndrome (high blood pressure, diabetes, high cholesterol, heart disease, and obesity) in comparison to the current medical care model (usual care) or providing healthy produce (medically tailored groceries).

DETAILED DESCRIPTION:
Many chronic conditions can be prevented, treated and improved, or even reversed through lifestyle modification. The practice and application of lifestyle medicine offers tremendous potential to restore health and reduce healthcare costs. Lifestyle Medicine is the use of evidence-based lifestyle therapeutic intervention-including a whole-food, plant-predominant eating pattern, regular physical activity, restorative sleep, stress management, avoidance of risky substances, and positive social connection-as a primary modality, delivered by clinicians trained and certified in this specialty to prevent, treat, and often reverse chronic disease. Lifestyle Medicine interventions have been applied in clinical, community, and workplace settings to drive health restoration and disease prevention.

In recent times there has been tremendous interest in the development and study of "Food Is Medicine" interventions as evidenced by the creation of a Food is Medicine initiative and inaugural Food is Medicine Summit, by the Department of Health and Human Services (HHS) in fiscal year 2023. Historically Food is Medicine interventions have been applied using 3 modalities:

Produce Prescriptions: Vouchers or restricted debit cards that can be redeemed for produce or direct distributions of produce that are made available to recipients based on a health condition or risk. Produce prescriptions are sometimes paired with services provided by RDNs, such as nutrition education, nutrition resources, supermarket tours, cooking classes, and medical nutrition therapy.

Medically Tailored Groceries: Distributions of unprepared or lightly processed foods that recipients are meant to prepare for consumption at home; the contents are sufficient to prepare nutritionally complete meals or provide a significant portion of the ingredients for such meals, including produce, whole grains and legumes, and lean proteins.

Medically Tailored Meals: Fully prepared meals made available through a referral from a medical professional or healthcare plan that are tailored to the medical needs of the recipient by a Registered Dietitian Nutritionist (RDN). Nutrition assessment, nutrition counseling and medical nutrition therapy are offered along with the meal program.

Food is medicine interventions suggest there is promise in improving not only food security, but health outcomes associated with diet related diseases. Addressing food insecurity with healthful food improving nutrition security is important, however "Food Is Medicine" interventions may not achieve the expected improvements in health outcomes if patient's lifestyle behaviors are not targeted comprehensively within their unique circumstances. This clinical aspect is often missing from the conversation in terms of chronic disease. Relative to "Food is Medicine" interventions, lifestyle medicine interventions are comprehensive expanding beyond nutrition, encompassing physical activity, stress management, smoking cessation, alcohol moderation, adequate sleep, and social connectivity to treat disease and drive health restoration.

The investigators research question is: Does a comprehensive lifestyle medicine intervention (involving culinary education, health education, physical activity, and urban agriculture) more effectively improve cardiometabolic risk factors in participants compared to those who only receive produce food boxes or usual care?

In a pilot pragmatic randomized control trial (pRCT), the investigators hypothesize that a comprehensive lifestyle medicine intervention can improve clinical outcomes (e.g., blood pressure, cholesterol levels, blood sugar levels, body mass index) of people are living with a lifestyle-related non-communicable disease such as obesity, heart disease, or diabetes compared to a medically tailored groceries cohort and usual care (acting as a control).

ELIGIBILITY:
Inclusion Criteria:

1. Cardiovascular Kidney Metabolic (CKM) syndrome as described by the American Heart Association (AHA)

   1. Stage 1 Metabolic Syndrome: Excess and/or dysfunctional adiposity

      * overweight/obesity - BMI ≥25 kg/m2 (or ≥23 kg/m2 if Asian ancestry)
      * abdominal obesity - Waist circumference ≥88/102 cm in women/men (or if Asian ancestry, ≥80/90 cm in women/men) and/or
      * dysfunctional adipose tissue
      * Fasting blood glucose ≥100-124 mg/dL or HbA1c between 5.7% and 6.4%*
      * without the presence of other metabolic risk factors or chronic kidney disease (CKD)
   2. Stage 2 Metabolic Syndrome: Metabolic risk factors and CKD

      * hypertriglyceridemia ≥135 mg/dL
      * hypertension
      * metabolic syndrome (MetS†)
      * waist circumference ≥88 cm for women and ≥102 cm for men (if Asian ancestry, ≥80 cm for women and ≥90 cm for men)
      * high-density cholesterol <40 mg/dL for men and <50 mg/dL for women
      * triglycerides ≥150 mg/dL
      * elevated blood pressure (BP) - systolic blood pressure ≥130 mm Hg and/or diastolic blood pressure ≥80 mm Hg and/or use of antihypertensive medications
      * fasting blood glucose ≥100 mg/dL
      * Diabetes (HbA1c > 6.5%)
      * CKD stage 1-3b
   3. Stage 3 Subclinical cardiovascular disease (CVD) in CKM

      * Risk equivalents of subclinical CVD- High predicted 10-y CVD risk
   4. Stage 4 Clinical CVD in CKM

      * Clinical CVD (coronary heart disease, heart failure, stroke, peripheral artery disease, atrial fibrillation) among individuals with excess/dysfunctional adiposity, other metabolic risk factors,
2. Electronic access to MyDataHelps platform either through an internet connected device like a personal computer, Ipad, or their personal phone and consent to its use
3. Must be patient of the NJ Family Practice Center at Rutgers Health/University Hospital

Exclusion Criteria:

1. Cardiovascular and Pulmonary Conditions

   * acute coronary syndrome with coronary artery bypass grafting in the past 3 months
   * uncontrolled hypertension with systolic BP > 160 or diastolic BP > 100
   * heart failure American College of Cardiology (ACC)/AHA Stage C and New York Heart Association (NYHA) > class II
   * life threatening or uncontrolled arrhythmia
   * hemodynamically relevant valvular heart disease
   * infiltrative heart disease including cardiac amyloidosis, sarcoidosis, Fabry's disease
   * genetic hypertrophic cardiomyopathy
   * significant pericardial disease
   * clinically significant congenital heart disease that may be cause of symptoms
   * significant anemia (hemoglobin <9)
   * severe chronic obstructive pulmonary disease (oxygen or steroid dependent)
   * severe restrictive pulmonary disease
2. Mental and Psychological Conditions

   * active suicidal behavior
   * substantial depressive symptoms. Antidepressant drugs are allowed if the dose has been stable for 3 months
   * uncontrolled major psychiatric illness (schizophrenia, bipolar, dementia)
   * history of drug or alcohol abuse or dependency within the past 12 months
   * history of medical noncompliance
   * Intellectual disability resulting in inability to make adult decisions
3. Musculoskeletal conditions

   * debility resulting in limited unassisted ambulation (being unable to walk 300 meters)
   * inability to perform activities of daily living unassisted
4. Other Major Organ System Conditions

   * very high-risk CKD (Stage 4 or 5 CKD or very high risk per Kidney Disease Improving Global Outcomes (KDIGO) classification)
   * significant hepatic dysfunction
   * untreated hypothyroidism or hyperthyroidism
   * cerebrovascular accident within past 6 months with functional residual deficits
   * clinically relevant neuromuscular disease
   * cancer or terminal illness with life expectancy < 3 years
   * pregnant or may become pregnant in the next 6 months
   * prior major organ transplant or intent to transplant (on the transplant list)
5. Administrative

   * participant in diabetes, nutrition, or weight research intervention in last 12 months
   * another family member or household member is a study participant. Only one member of each household may take part in this study.
   * individuals who have started treatment with a class of medications known as GLP-1 within 120 days of the program start
   * individuals who have undergone bariatric surgery.
   * participants without smartphone or web access
   * individuals who are not proficient in English to a level that would allow for unassisted understanding of study materials and informed consent documentation, as well as effective communication with the research team
   * individuals currently facing acute unresolved health-related social needs, including but not limited to, unstable housing, lack of reliable transportation, and unemployment
   * These conditions are considered exclusion criteria due to the potential for it to significantly impact their ability to participate consistently in the study. It can affect the individual's ability to adhere to study protocols, attend follow-up appointments, or impact the generalizability of the study findings. The investigators recognize the importance of addressing these social determinants of health, typically in clinical practice the investigators focus on helping the patient stabilize and resolve health related social needs prior to engaging in a comprehensive therapeutic lifestyle change program.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Disease reversal | 12 weeks after start of intervention
  Reduction of disease measures below the threshold for diagnosing the target disease/condition with an absence of medications or procedures known to affect those measures.
Medication reduction | 12 weeks after start of intervention
  A decrease in the prescribed dose to the next appropriate dose of a specific agent for a specific condition

SECONDARY OUTCOMES:
Food Security | 12 weeks after start of intervention
  Defined as access by all members, at all times to have enough food for an active, healthy life
Diet Quality | 12 weeks after start of intervention
  Diet quality is broadly defined as a dietary pattern or an indicator of variety across key food groups relative to those recommended in dietary guidelines. Diet quality is objectively measured using the Healthy Eating Index (HEI) 2020
Culinary Attitudes and Behaviors | 12 weeks after start of intervention
  Assessed using the "Cooking With A Chef" survey instrument which consists of 8 scales assessing: 1. availability and accessibility of fruits and vegetables (AAFV), 2. cooking attitudes (CA) 3. cooking behaviors (CB), 4. produce consumption self efficacy (SEPC) , 5. cooking self-efficacy (SEC), 6. self-efficacy for using basic cooking techniques (SECT) and 7. self-efficacy for using fruit, vegetables, and seasonings (SEFVS) 8. knowledge of cooking terms and techniques.
Physical Activity | 12 weeks after start of intervention
  Self-reported and measured duration and intensity of physical activity

OTHER OUTCOMES:
Hemoglobin A1C | 12 weeks after start of intervention
  Measure of glycosylated hemoglobin and diagnostic test for diabetes
Maximum Oxygen Uptake (VO2 Max) | 12 weeks after start of intervention
  Estimated amount of oxygen uptake possible measured by the YMCA step test.
Total Body Strength as measured by the Isometric Mid-Thigh Pull | 12 weeks after start of intervention
  Quantitative test of total body strength using an instrumented dead lift technique measured in Newtons of force per kilogram of body weight.
Waist Circumference | 12 weeks after start of intervention
  a surrogate measure of visceral adiposity and one component of metabolic syndrome
Waist to Hip Ratio | 12 weeks after intervention start
  waist circumference measurement divided by the hip circumference measurement. Ratio used to assess non-communicable disease risk
Low-Density Lipoprotein Cholesterol (LDL-C) | 12 weeks after intervention start
  diagnostic laboratory test assessing low-density lipoprotein cholesterol concentration that correlates with cardiovascular disease risk
Blood Pressure | 12 weeks after intervention start
  Measurement of arterial wall pressure and risk factor for cardiovascular disease
Grip Strength | 12 weeks after intervention start
  A simple and reliable measurement of maximum voluntary muscle strength derived from combined contraction of extrinsic and intrinsic hand muscles
Body Weight | 12 weeks after intervention start
  The mass or quantity of heaviness of an individual, expressed by units of pounds or kilograms
Perceived Program Impact | 12 weeks after intervention start
  Assessed using "Most Significant Change" tool. It is a qualitative survey tool that assesses an individual's perspective on what caused the most significant change associated with an intervention and why.
Non High-Density Lipoprotein Cholesterol (Non-HDL-C) | 12 weeks after intervention start
  measure of all atherogenic lipoproteins and cholesterol, including low-density lipoprotein (LDL) but excludes high density lipoprotein (HDL)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lynch, PT, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers Health New Jersey Family Practice Center, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT06461273/ICF_000.pdf